CLINICAL TRIAL: NCT00620802
Title: A Phase I, Open-Label, Randomized, Multiple-Dose, Two-Way Crossover Study of the Pharmacodynamics of CGT 2168 Compared With Plavix®
Brief Title: Pharmacodynamics of CGT 2168 Compared With Plavix®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cogentus Pharmaceuticals (Industry)
Responsible Party: Pablo Lapuerta, MD, Cogentus Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CG106
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: Platelet function testing; Healthy volunteers
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): CGT-2168 (clopidogrel 75 mg/omeprazole 20 mg)
  Interventions: Drug: CGT-2168
- B (Active Comparator): Plavix (clopidogrel 75 mg)
  Interventions: Drug: Plavix

INTERVENTIONS:
Drug: CGT-2168 — (CGT-2168, one capsule each daily)
  Arms: A
Drug: Plavix — (clopidogrel, 75 mg)
  Arms: B

SUMMARY:
CG106 is a Phase I open-label, randomized, multiple-dose, two-way crossover study to characterize the pharmacodynamics and pharmacokinetics of the investigational fixed-dose combination product CGT 2168 (clopidogrel, 75 mg and omeprazole, 20 mg) relative to Plavix® (clopidogrel, 75 mg).

Healthy volunteer subjects will undergo two dosing periods. In each 7-day dosing period, subjects will receive oral doses of study drug consisting of open-label CGT 2168 or Plavix® in the order determined by the randomization schedule. Each period of dose administration will be separated by a two-week washout period. Study exit will occur 1 week after Dosing Period 2. The expected total duration of participation is 8 weeks (56 days), including a screening visit on or within 21 days prior to enrollment.

On the day before Day 1 and Day 7 in each dosing period, subjects will be admitted to the Phase I unit. Blood samples to determine ADP-induced platelet aggregation will be collected pre-dose on Day 1 and 2 h after dosing on Day 7. Plasma concentrations of clopidogrel parent and clopidogrel carboxylic acid metabolite will also be measured pre-dose on Day 1 and pre-dose and serially after dosing on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females. Women of childbearing potential must have a negative pregnancy test prior to enrollment and agree to use two methods of effective barrier contraception, or a hormonal contraceptive to prevent pregnancy throughout the study.
* Able to comply with study procedures, which includes returning to the Phase I unit for all scheduled visits and procedures.
* Abstinence from tobacco use (including smoking cessation products containing nicotine) for 90 days prior to study entry, with agreement to abstain from tobacco/nicotine use throughout the study.
* Agreement to abstain from alcohol and caffeine ingestion from 72 h before dosing and throughout each dosing period.
* Able to give informed consent, and subject has signed and dated a written consent form approved by the IRB.

Exclusion Criteria:

* Hypersensitivity to clopidogrel, omeprazole, or related drugs including inactive ingredients.
* BMI (body mass index) outside the range of 19-30 kg/m2.
* At screening, body weight less than 50 kg if male or 45 kg if female.
* Clinically significant abnormal findings on physical examination, clinical laboratory tests or ECG at screening.
* History of hypertension or 5-minute sitting screening BP ≥160/100 mmHg on measurements repeated twice.
* History of diabetes mellitus, renal failure, acute or chronic liver disease, including acute or chronic hepatitis, or cirrhosis.
* Positive HIV-1 antibody, hepatitis B surface antigen or hepatitis C antibody screening test.
* History of any clinically significant medical or psychiatric condition.
* Difficulty in swallowing medication, or any known or suspected gastrointestinal abnormality that may affect drug absorption.
* Participation in a previous clinical trial within 30 days prior to enrollment (check-in on Day -1 for Visit 2).
* Blood donation of ≥ 1 pint within 30 days or plasma donation within 14 days prior to enrollment (check-in on Day -1 for Visit 2).
* Use of any prescription or over-the-counter medications or ingestion of herbal drugs/dietary supplements including vitamins and minerals within 14 days prior to enrollment (check-in on Day -1 for Visit 2). Hormonal contraceptives are allowed.
* Subject is not willing to refrain from drinking grapefruit juice or eating grapefruit throughout study participation.
* Subject is an active illicit drug user or has a history of illicit drug use within the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is inhibition of platelet aggregation (IPA) based on maximum platelet aggregation (MPA) to 5 and 20 µM ADP after 7 days daily dosing with CGT-2168 compared to Plavix®. | 7 days

SECONDARY OUTCOMES:
Residual aggregation, measured 10 min after the addition of 20 and 5 µM ADP, after 7 days daily dosing with CGT 2168 compared to Plavix®. | 7 days
Plasma PK measures of clopidogrel (parent drug and carboxylic acid metabolite) with CGT 2168 compared to Plavix®. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lapuerta, MD, Study Director — Cogentus Pharmaceuticals
Locations (1):
- Quintiles Phase I Services, Overland Park, Kansas, United States